CLINICAL TRIAL: NCT00912977
Title: Prospective Evaluation of Forceplate Measured Levodopa-Induced Dyskinesia
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kathryn Anne Chung, Associate Professor, Oregon Health and Science University
Other Study IDs: e5348
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinsons disease; dyskinesia; measurement
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Groups are defined by another study
- Group 2: Groups are defined by another study
- Group 3: Groups are defined by another study

SUMMARY:
Nearly all Parkinson's disease (PD) patients eventually develop abnormal and unwanted movements (dyskinesias; LID) caused by the gold standard treatment, Levodopa. The severity of these movements can range from subtle to extremely debilitating and may or may not interfere with normal activities such as putting on a coat or brushing ones teeth. The purpose of this study is to demonstrate the validity and reliability of objectively measuring dyskinesia with a forceplate.

DETAILED DESCRIPTION:
The main outcome measure of this study are measurements taken every half hour during an inpatient study visit. These measurements include standing on a forceplate for 1 minute while performing a mental task such as reciting the alphabet backwards. During this forceplate stance, a rater will visually score your movements. All participants must be eligible for another Parkinson's disease study at Oregon Health and Science University.

ELIGIBILITY:
Inclusion Criteria:

* Parkinsons disease
* Older than 18

Exclusion Criteria:

* Must be participating in a Parkinsons disease study at Oregon Health & Science University

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinsons disease patients with levodopa-induced dyskinesia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Forceplate Measure | Every 1/2 hour

SECONDARY OUTCOMES:
Visual Rating Scale | every 1/2 hour

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Chung, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Durif F, Debilly B, Galitzky M, Morand D, Viallet F, Borg M, Thobois S, Broussolle E, Rascol O. Clozapine improves dyskinesias in Parkinson disease: a double-blind, placebo-controlled study. Neurology. 2004 Feb 10;62(3):381-8. doi: 10.1212/01.wnl.0000110317.52453.6c. PMID 14872017
- [Background] Hagell P, Widner H. Clinical rating of dyskinesias in Parkinson's disease: use and reliability of a new rating scale. Mov Disord. 1999 May;14(3):448-55. doi: 10.1002/1531-8257(199905)14:33.0.co;2-0. PMID 10348468
- [Background] Durif F, Vidailhet M, Debilly B, Agid Y. Worsening of levodopa-induced dyskinesias by motor and mental tasks. Mov Disord. 1999 Mar;14(2):242-5. doi: 10.1002/1531-8257(199903)14:23.0.co;2-w. PMID 10091616